CLINICAL TRIAL: NCT06860555
Title: Exploration of the Retinal Deep PhenotypingTM (RDP) Platform for the Identification of Spatial-spectral Features in Different Types of Drusenoid Deposits in Dry Age-related Macular Degeneration (AMD)
Brief Title: Hyperspectral Drusen Classification
Status: Completed | Type: Observational
Sponsor: Optina Diagnostics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 22-003
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Dry Age Related Macular Degeneration
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Participants with dry AMD: Participants with dry AMD in at least one eye will undergo a hyperspectral retinal imaging session with Optina Diagnostics' MHRC in addition to retinal imaging with OCT, used as the gold standard method to identify and classify the drusenoid deposits.
  Interventions: Device: Mydriatic Hyperspectral retinal Camera, (MHRC) and Optical coherence tomography (OCT)

INTERVENTIONS:
Device: Mydriatic Hyperspectral retinal Camera, (MHRC) and Optical coherence tomography (OCT) — Imaging with the MHRC and optical coherence tomography (OCT).

SUMMARY:
This observational, cross-sectional study is designed to explore the feasibility to extract spatial-spectral features from hyperspectral retinal images captured with Optina Diagnostics' MHRC that are characteristic to the different types of drusenoid deposits associated with dry age-related macular degeneration.

DETAILED DESCRIPTION:
In this observational, cross-sectional, prospective study, participants with dry AMD in at least one eye will undergo a hyperspectral retinal imaging session with the Optina Diagnostics' MHRC in addition to retinal imaging with OCT, used as the gold standard method to identify and classify the drusenoid deposits.

Eligible participants visiting the eye clinic for AMD with dry AMD in at least one eye will be invited to participate in the study. Subjects who sign an informed consent to participate in the study will have their eyes evaluated to confirm that at least one eye is meeting all of the inclusion criteria, and none of the exclusion criteria. The dry AMD status and stage as well as information about eye diseases and conditions will be documented for both eyes. If eligible (no ocular exclusion criteria present in at least one eye), subjects will undergo OCT imaging of the macular region. If the OCT imaging session is successful (as described in the OCT imaging procedure below), the participants will then undergo hyperspectral retinal imaging with the Optina Diagnostics MHRC.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for participation, volunteers must conform to all of the following inclusion criteria:

  * Male and female adults aged 50 years and older (inclusive).
  * Dry AMD in at least one eye, with at least one type of the following retinal drusenoid deposits: reticular pseudodrusen, soft drusen, hard drusen.

    ○ The presence of multiple small drusen (< 63µm) or intermediate drusen (≥63µm and ≥125µm) is sufficient to qualify for this study (Coleman, 2008).
  * Ability and willingness to give informed consent.

Exclusion Criteria:

Individuals that meet any of the following exclusionary criteria cannot be enrolled:

* Any ophthalmologic condition that would prevent obtaining retinal imaging and/or could interfere with the analysis of the MHRC images and OCT images, including:

  * Pupil dilation contraindicated (due to a pathology or with 3 quadrants with Van Herick of 0 or 1 without iridotomy)
  * Inadequate pupil dilatation (< 6mm diameter) preventing uniform illumination of the retina with the MHRC
  * Dry AMD presenting only with pigmentary changes or geographic atrophy (no drusenoid deposits)
  * Presence of geographic atrophy in a cumulative area of >0.5 disc area
  * Presence of neovascular AMD, defined as the presence of at least 1 of the following 4 characteristics: serous sensory retinal detachment, RPE detachment, subretinal hemorrhage, or subretinal fibrous tissue; or history of photocoagulation for choroidal new vessels (AREDS, 2005)
  * Signs of vascular occlusion or retinopathy (microaneurysm, exudate, hemorrhage or edema) within a diameter of 10 mm from the mid-point between the optic nerve head and the macula (i.e. the area of interest for the MHRC imaging)
  * Macular dystrophy
  * Nuclear sclerosis > 2 (LOCS II four-point grading system) or presence of central cortical or central posterior subcapsular cataract
  * Deficient visual fixation (inability to fixate for at least 2 s)
  * Refractive error outside the range of -15 D to +15 D
  * Corneal or media opacities (e.g. Weiss ring) affecting retinal imaging on a cumulative area > 1 disc area within a diameter of 10 mm from the mid-point between the optic nerve head and the macula (i.e. the area of interest for the MHRC imaging)
  * Scar, atrophy, naevus, tumor, epiretinal membrane or retinal pucker with a cumulative area > 1 disc area within a diameter of 10 mm from the mid-point between the optic nerve head and the macula (i.e. the area of interest for the MHRC imaging).
  * Papilledema
* Inability to obtain an OCT image centered on the macular region of satisfactory quality for analysis of the drusenoid deposits (as indicated by the OCT's software quality indicator)
* Inability of obtaining at least 3 images of satisfactory quality with the MHRC per the Optina Diagnostics quality index software.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 50 years old and above with dry AMD with the presence of drusenoid deposits in at least one eye.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Creation of a bank of hyperspectral retinal images | 12 months
  Creation of a bank of hyperspectral retinal images that are normalized, registered, segmented and annotated by visual inspection for drusenoid deposit types (soft, hard or reticular pseudodrusen) identified in OCT images re-examined in these re
Evaluation of the segmented drusenoid deposit | 12 months
  Evaluation of the segmented drusenoid deposit to identify characteristic spatial-spectral features extracted with the use of a method such as, but not limited, to spatial-spectral texture analysis, local spectral normalization, spectral angle mapper (SAM) or Dimension Reduction by Orthogonal Projection for Discrimination (DROP-D) for each type and a creation of classifier.
Explore if spatial-spectral features identified for different drusenoid deposit | 12 months
  Explore if spatial-spectral features identified for different drusenoid deposit types, and in particular for soft drusen, may be present in locations outside the segmented regions visible to the observer on the hyperspectral images and OCT images. Indeed, these regions could be related to basal linear and basal laminar deposits regions and the OCT scans could be re-examined in these regions to evaluate if there is a visible "split" between the RPE and Bruch's membrane previously associated with basal laminar deposits (Sura et al., 2020).
Effect of the location each type of drusenoid deposit | 12 months
  Explore the effect of the location each type of drusenoid deposit on the characteristic spatial-spectral features. In this optional sub-study, the drusenoid deposit annotations will include the location based, for example, on circles centered on the fovea within a diameter of 1 mm, 3 mm, 6 mm and beyond 6 mm (if available in the OCT images). (Optional)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jean Daniel Arbour, MD, FRCSC, Principal Investigator — Clinique Ophtalmologique 2121, 2121 rue Sherbrooke Ouest, Montréal, Québec, H3H 1G6
Locations (1):
- Clinique Ophtalmologique 2121, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No